CLINICAL TRIAL: NCT06734988
Title: Japanese Esophageal Pressure Sub-study of EXTubation Evaluation and Respiratory Dynamics in Acute Respiratory Distress Syndrome (EXTEND ARDS-J EP Study)
Brief Title: EXTEND ARDS-J Esophageal Pressure Study
Status: Recruiting | Type: Observational
Sponsor: Sapporo Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: EXTEND_ARDS_J_EP_Study
Record Dates: First submitted 2024-12-04; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
Keywords: Esophageal pressure; SBT
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mechanically ventilated adult ARDS patients: Adult mechanically ventilated patients (≥ 16 years old) with esophageal pressure monitoring, expected to receive invasive mechanical ventilator for more than 48 hours

SUMMARY:
Background: Acute respiratory distress syndrome (ARDS) patients require careful assessment before extubation to prevent failure, which is associated with poor outcomes. While current guidelines recommend weaning protocols, these are based on general respiratory failure studies rather than ARDS-specific data. Esophageal pressure (Pes) measurement provides direct assessment of inspiratory effort but is rarely utilized clinically.

Objectives: This Japanese sub-study of EXTEND ARDS aims to evaluate whether:

1. ΔPes measurements during spontaneous breathing trials (SBT) can predict SBT failure
2. ΔPes measurements post-extubation can predict 48-hour extubation failure

Methods: This prospective observational study will be conducted in Japanese ICUs. Esophageal pressure will be measured using standardized Nutrivent balloons (4mL volume) with Hamilton ventilators. Balloon placement in the lower third of the esophagus will be confirmed by cardiac artifacts and chest X-ray. ΔPes will be calculated as the difference between end-expiratory and peak inspiratory esophageal pressure, excluding esophageal contractions.

Significance: This study addresses a knowledge gap regarding the utility of esophageal pressure monitoring in ARDS patients during mechanical ventilation weaning. Findings may help optimize extubation timing and improve patient outcomes through objective physiological measurements.

DETAILED DESCRIPTION:
1. Background Acute respiratory distress syndrome (ARDS) remains a life-threatening condition with high mortality among mechanically ventilated patients. While current guidelines recommend weaning protocols for extubation, these are primarily based on studies of general acute respiratory failure rather than ARDS-specific populations.

   Inspiratory effort assessment during liberation from mechanical ventilation traditionally relies on respiratory rate monitoring during spontaneous breathing trials (SBT). However, esophageal pressure (Pes) measurement, which provides direct measurement of inspiratory effort, is rarely utilized in clinical practice. This is particularly relevant in ARDS patients, where excessive inspiratory effort can induce pendelluft phenomenon, potentially causing dorsal lung injury in the supine position.

   Recent studies have shown that diaphragmatic contraction, maximum inspiratory pressure, ΔPes, and trans-diaphragmatic pressure can predict successful weaning in prolonged mechanical ventilation patients. However, there remains a significant knowledge gap regarding the utility of esophageal pressure measurements in predicting SBT and extubation success specifically in ARDS patients.
2. Study Significance This Japanese sub-study of the EXTEND ARDS trial will investigate whether ΔPes measurements during SBT and post-extubation can predict extubation outcomes in ARDS patients. By incorporating esophageal pressure monitoring, this study aims to provide objective physiological data to improve the prediction of extubation success and optimize the timing of liberation from mechanical ventilation.
3. Study Design and Methods This is a prospective observational sub-study conducted in Japanese ICUs. Esophageal pressure will be measured using Nutrivent balloons with Hamilton C6 or G5 ventilators. The balloon placement will be confirmed by cardiac artifacts and chest X-ray, positioned in the lower third of the esophagus. Balloon volume will be standardized at 4mL, following manufacturer recommendations and GLOBAL WEAN study protocols.
4. Primary Objectives

To evaluate whether:

1. ΔPes measurements during SBT can predict SBT failure
2. ΔPes measurements post-extubation can predict extubation failure within 48 hours

ELIGIBILITY:
Inclusion Criteria:

1. Adult mechanically ventilated patients (≥ 16 years old) with esophageal pressure monitoring, expected to receive invasive mechanical ventilator for more than 48 hours
2. Patients who meet the diagnosis of ARDS at the start of invasive mechanical ventilation based on a new global definition of ARDS.

Exclusion Criteria:

1. Patients who already had tracheostomy at the start of invasive mechanical ventilation
2. Patients who were transferred to participating hospital more than 2 days after the start of invasive mechanical ventilation
3. Patients with terminal conditions at the start of invasive mechanical ventilation
4. Patients who have expressed their refusal to have their clinical data used in research

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult mechanically ventilated patients (≥ 16 years old) expected to receive invasive mechanical ventilator for more than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Reintubation within 48 hours after extubation | 48 hours after extubation
  Occurrence of reintubation events within 48 hours after planned extubation

SECONDARY OUTCOMES:
SBT Failure | Up to 120 minutes from the start of spontaneous breathing trial
  Occurrence of SBT failure defined as inability to complete the spontaneous breathing trial

OTHER OUTCOMES:
90 days in-hospital mortality | From intubation to 90 days after intubation
  90 days in-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Sapporo Medical University, Sapporo, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol